CLINICAL TRIAL: NCT03768518
Title: The Physiology of Glucagon-like-peptide-1 Espression in Patients With Endogenous Hyperinsulinism: Correlation With Histopathology
Brief Title: GLP-1 Receptor Expression in CHI
Acronym: GLP-1-CHI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: European Commission (Other); University College, London (Other); Charite University, Berlin, Germany (Other); University Hospital, Basel, Switzerland (Other); Insel Gruppe AG, University Hospital Bern (Other); University of Helsinki (Other); Turku University Hospital (Other Government); University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Martin Gotthardt, Professor, Radboud University Medical Center
Other Study IDs: NL54275.091.15
Record Dates: First submitted 2018-07-11; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Congenital Hyperinsulinism
Keywords: Exendin; GLP-1; PET/CT
MeSH Terms: conditions — Congenital Hyperinsulinism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 68Ga-exendin-4 PET/CT — 68Ga-exendin-4 PET/CT

SUMMARY:
The primary objective is the in vivo and ex vivo investigation of the expression and distribution of the GLP-1R in the pancreas of CHI patients.

DETAILED DESCRIPTION:
Congenital hyperinsulinism (CHI) is a rare disease of infants characterized by the presence of functionally defective non-neoplastic beta-cells with inappropriate (over-) secretion of insulin, leading to life-threatening hypoglycaemia. Beta cells specifically express the glucagon-like-peptide-1 (GLP-1R), which could be a promising target for diagnostic and therapeutic purposes. In this study we propose to investigate the physiology of GLP-1 receptor expression in CHI. Expression of the GLP-1 receptor will be quantified in vivo by 68Ga-NODAGA-exendin-4 PET/CT. This data will be compared with post-surgical autoradiography and morphometric determinations.

Furthermore, we will evaluate 68Ga-exendin-4 PET/CT for the pre-operative localization of foci of over-secreting beta cells in CHI and the discrimination between focal and diffuse CHI. We will compare GLP-1R PET/CT to the currently used pre-operative imaging technique (18F-DOPA PET combined with contrast enhanced CT). To compare these imaging techniques according to sensitivity, we will analyze intra-operative findings and clinical outcomes.

These highly relevant data will allow us to evaluate the expression of GLP-1R in CHI and its usefulness as a target for diagnosis of this disease. Since the localization of foci in CHI and the discrimination between focal and diffuse CHI is challenging, surgical removal of unnecessary large portions of the pancreas in frequently necessary. Evaluation of a better target for pre-operative imaging would therefore be of great value.

Objective:

The primary objective is the in vivo and ex vivo investigation of the expression and distribution of the GLP-1R in the pancreas of CHI patients. A 68Ga-NODAGA-exendin 4 PET/CT will be performed in all patients included in this study. The results of quantitative imaging will then be compared to GLP-1R expression and autoradiography of surgical specimens to determine the interdependency of radiotracer uptake, beta cell mass and GLP-1R expression.

Furthermore, GLP-1R imaging will be compared to the standard imaging techniques now used in pre-operative imaging of children with CHI. All patients will undergo the standard imaging procedure, consisting of an 18F-DOPA PET scan combined with a contrast-enhanced CT. The results of the GLP-1R imaging will be compared to standard imaging in respect to sensitivity for localization of the lesion and discrimination between focal and diffuse CHI. This will be determined by the comparison of the results of pre-operative imaging with intra-operative findings.

Also, the safety (side-effects) of 68Ga-NODAGA-exendin and 18F-DOPA will be assessed.

Furthermore, dosimetric calculations will be performed and the minimum radioactivity dose of 68Ga-NODAGA-exendin 4 to obtain acceptable/reliable images will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Biochemically and clinically proven endogenous congenital hyperinsulinism:
* Unresponsive to medical treatment (diazoxide)
* Indication for 18F-DOPA PET/CT based on mutation analysis
* Standard imaging (18F-DOPA PET/CT) not older than 8 weeks
* <16 years old
* Informed consent signed by parents or legal guardians of the patient.

Exclusion Criteria:

* Genetically proven diffuse CHI (presenting with a homozygous or compound heterozygous ABCC8/KCNJ11 mutation)
* Calculated creatinine clearance below 40 ml/min
* Evidence of other malignancy than insulin producing tumors in conventional imaging (suspicious liver, bone and lung lesions based on CT)
* Age > 16 years
* No signed informed consent

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients (<16 years) with biochemically proven endogenous congenital hyperinsulinism
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-02-07 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Expression and distribution of GLP-1R in pancreas of children with CHI | 1 year
  Comparison of PET quantification with autoradiography and histology

SECONDARY OUTCOMES:
Comparison of the exendin PET/CT and F-DOPA PET/CT | 1 year
  Comparison of sensitivity and specificity for localization of focal CHI

CONTACTS AND LOCATIONS:
Overall Officials: Martin Gotthardt, Prof., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands